CLINICAL TRIAL: NCT02506231
Title: The Effect of Folinic Acid Rescue Following Methotrexate (MTX) Graft-versus-host Disease (GVHD) Prophylaxis on Regimen Related Toxicity and Transplantation Outcome: a Double Blind Randomized Controlled Study
Brief Title: The Effect of Folinic Acid Rescue Following MTX GVHD Prophylaxis on Regimen Related Toxicity and Transplantation Outcome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0197-15-RMC
Record Dates: First submitted 2015-07-13; First posted 2015-07-23 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-06

CONDITIONS: Graft vs Host Disease; Allogeneic Hematopoietic Cell Transplantation; Mucositis
Keywords: Allogeneic hematopoietic cell transplantation; GVHD prophylaxis; Methotrexate; Folinic acid; Leucovorin; Mucositis
MeSH Terms: conditions — Graft vs Host Disease; Mucositis | interventions — Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Folinic acid (Experimental): Patients will be randomly assigned by central randomization in a 1:1 ratio to receive folinic acid (FA) or placebo starting 24h after each MTX dose for 24h. Oral FA 15 mg/dose or placebo will be given every 8h after MTX administration on day 1 (3 doses), and every 6h (4 doses) on days 3 and 6.
  Interventions: Drug: Folinic acid
- Placebo (Placebo Comparator): Patients will be randomly assigned by central randomization in a 1:1 ratio to receive folinic acid (FA) or placebo starting 24h after each MTX dose for 24h. Oral FA 15 mg/dose or placebo will be given every 8h after MTX administration on day 1 (3 doses), and every 6h (4 doses) on days 3 and 6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Folinic acid
  Other Names: leucovorin
  Arms: Folinic acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the impact of folinic acid (FA) -rescue following methotrexate (MTX) graft-versus-host disease (GVHD) prophylaxis on regimen related toxicity and transplantation outcomes after allogeneic hematopoietic cell transplantation (alloHCT) in a double blind randomized controlled trial.

DETAILED DESCRIPTION:
A regimen consisted on a combination of a calcineurin inhibitor (CNI) with a short course of methotrexate (MTX) is the most widely used regimen for the prevention of GVHD after allogeneic hematopoietic cell transplantation (alloHCT). While the CNI is given in an adjusted dose, based on blood levels, MTX is given at a fixed 3 or 4 doses (15 mg/m2 on day +1, 10 mg/m2 on days +3, +6 +/- day +11). However, its use may be associated with considerable toxicity, including delayed engraftment, hepatotoxicity, nephrotoxicity and particularly oral mucositis (OM). The basis for OM is integrated: conditioning regimen and MTX prophylaxis for acute GVHD. OM has been shown to be associated with increased mortality and morbidity (principally from infection), significant pain, dysgeusia, difficulty speaking, difficulty receiving nutrition, hydration and oral medications, prolonged hospitalization and increased costs of care.

Reducing and even omitting doses of MTX due to regimen related toxicities (mucositis, hepatic and renal toxicities) is common. However, dose reduction of MTX may be associated with increased risk of acute GVHD and early death. Several non-randomized studies have shown that folinic acid (FA, leucovorin) administration may reduce MTX toxicity. Nevertheless, the efficacy and safety of its administration remain controversial. Despite limited and uncontrolled data, the European Group for Blood and Marrow Transplantation (EBMT) and the European LeukemiaNet working group recently recommended the use of FA-rescue and proposed a uniform policy of FA-rescue 24h after each MTX dose: 15mg every 8h after MTX administration on day 1, and every 6h on days 3, 6 and 11. Yet, according to several surveys (including by EBMT-ELN) only half of bone marrow transplantation (BMT) centers use to give post MTX FA-rescue.

The aim of this study is to assess the impact of FA-rescue following MTX GVHD prophylaxis on regimen related toxicity and transplantation outcomes after alloHCT in a double blind randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute leukemia in complete remission (CR) or myelodysplastic syndrome;
* First transplantation;
* Peripheral blood graft;
* Matched sibling or unrelated donor or one antigen or allelic mismatched sibling or unrelated donor (10/10 or 9/10 human leukocyte antigen match );
* Myeloablative or reduced intensity preparative regimen;
* Post-transplant GVHD prophylaxis consisting of a calcineurin inhibitor (CSA or tacrolimus) and methotrexate;
* Glutamate Pyruvate Transaminase (GPT) < 3 times upper normal limit (UNL) and creatinine ≤ 1.4 mg%;
* Written informed consent;

Exclusion Criteria:

* True non-myeloablative preparative regimen (TBI 200 +/- fludarabine);
* Acute leukemia not in remission;
* GPT > 3 times upper normal limit or creatinine > 1.4 mg%;
* Bone marrow, haploidentical or cord blood grafts;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe (grade 3-4) oral mucositis according to the WHO scale | 30 days
  According to the WHO (world health organization) oral mucositis grading scale
Duration (in days) of severe (grade 3-4) oral mucositis according to the WHO scale | 30 days
  According to the WHO (world health organization) oral mucositis grading scale

SECONDARY OUTCOMES:
Incidence of oral mucositis | 30 days
Grade of oral mucositis | 30 days
  According to the WHO (world health organization) oral mucositis grading scale
Time to neutrophil recovery | 30 days
Time to platelet recovery | 60 days
Adherence to methotrexate schedule | 14 days
  Number of methotrexate doses that were actually given (out of 3 doses on days 1, 3 and 6)
Adherence to methotrexate doses | 14 days
  Actual methotrexate doses given in mg/sqm divided by scheduled doses in mg/sqm X 100
Days of opiate use | 30 days
Days of total parenteral nutrition use | 100 days
Incidence of veno-occlusive disease of the liver (VOD) | 30 days
Severity of veno-occlusive disease of the liver (VOD) | 30 days
  According to the Seattle criteria
Incidence of renal toxicity | 30 days
  Creatinine > 2 mg%
Incidence of hepatic toxicity | 30 days
  total bilirubin > 2 mg%, unless mostly indirect
Incidence of febrile neutropenia | 30 days
Duration of febrile neutropenia | 30 days
Documented infections | 30 days
Time from transplantation to discharge | 60 days
Incidence of acute graft-versus-host disease | 100 days
Severity of acute graft-versus-host disease | 100 days
  According to the consensus grading system
Incidence of chronic graft-versus-host disease | 24 months
Severity of chronic graft-versus-host disease | 24 months
  According to the National Institutes of Health (NIH) consensus criteria
Incidence of relapse | 24 months
Non relapse mortality | 24 months
Disease free survival | 24 months
Overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Yeshurun, MD, Principal Investigator — Rabin Medical Center

REFERENCES:
- [Derived] Yeshurun M, Rozovski U, Pasvolsky O, Wolach O, Ram R, Amit O, Zuckerman T, Pek A, Rubinstein M, Sela-Navon M, Raanani P, Shargian-Alon L. Efficacy of folinic acid rescue following MTX GVHD prophylaxis: results of a double-blind, randomized, controlled study. Blood Adv. 2020 Aug 25;4(16):3822-3828. doi: 10.1182/bloodadvances.2020002039. PMID 32790844